CLINICAL TRIAL: NCT00002170
Title: A Pilot, Phase II, Randomized, Placebo-Controlled Study to Determine the Effects of Viracept on the Clinical Outcome of Disseminated Mycobacterium Avium Complex Disease (MAC) in AIDS Patients Who Are Receiving Standard Acute Treatment for This Opportunistic Infection
Brief Title: A Study of Viracept in AIDS Patients With Mycobacterium Avium Complex Disease (MAC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Agouron Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 259C; Study 518; AG1343-518
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-05

CONDITIONS: Mycobacterium Avium-Intracellulare Infection; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Placebos; Mycobacterium avium-intracellulare Infection; Acquired Immunodeficiency Syndrome; HIV Protease Inhibitors; Nelfinavir; Anti-Infective Agents; Anti-HIV Agents
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — Nelfinavir

INTERVENTIONS:
Drug: Nelfinavir mesylate

SUMMARY:
The purpose of this study is to see if it is safe and effective to give Viracept to AIDS patients who are being treated for MAC.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV infection
* New diagnosis of MAC bacteremia and < 7 days of therapy.

Prior Medication:

Allowed:

Patients no more than 7 days of therapy for MAC disease.

Exclusion Criteria

Prior Medication:

Excluded:

Prior therapy (or less than 2 weeks) with protease inhibitors other than saquinavir.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - Harbor UCLA Med Ctr, Torrance, California
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Boston VA Med Ctr / 151, Boston, Massachusetts
  - Baylor Univ, Houston, Texas